CLINICAL TRIAL: NCT04082975
Title: A Randomized, Double-blind, Active Controlled, Parallel, Multicenter, Phase 3 Clinical Trial to Evaluate the Efficacy and Safety of NVP-1203 in Patients With Acute Low Back Pain
Brief Title: Efficacy and Safety of NVP-1203 and NVP-1203-R in Patients With Acute Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: NVP Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NVP-1203_P3
Record Dates: First submitted 2019-09-04; First posted 2019-09-10 (Actual); Last update posted 2021-06-07 (Actual); Status verified 2021-06

CONDITIONS: Acute Low Back Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NVP-1203 (Experimental): NVP-1203 plus NVP-1203-R placebo for up to 7 days, oral dose
  Interventions: Drug: NVP-1203; Drug: NVP-1203-R placebo
- NVP-1203-R (Active Comparator): NVP-1203-R plus NVP-1203 placebo for up to 7 days, oral dose
  Interventions: Drug: NVP-1203-R; Drug: NVP-1203 placebo

INTERVENTIONS:
Drug: NVP-1203 — Oral dose for 7 days
  Arms: NVP-1203
Drug: NVP-1203-R — Oral dose for 7 days
  Arms: NVP-1203-R
Drug: NVP-1203 placebo — Oral dose for 7 days
  Arms: NVP-1203-R
Drug: NVP-1203-R placebo — Oral dose for 7 days
  Arms: NVP-1203

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety NVP-1203 in patients with acute low back pain.

DETAILED DESCRIPTION:
This study is a randomized, double-blind, active-controlled, parallel, phase 3 study to evaluate efficacy and safety of NVP-1203 in patients with acute low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have ability to comprehend the contents of study and before participating in trial and have willingness to sign of informed consent in writing
* Subjects who have symptom of acute low back pain

Exclusion Criteria:

* Subjects who cannot prohibit anti-inflammatory drug or muscle relaxants during clinical trial
* Inadequate subject for the clinical trial by the investigator's decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 421 (Actual)
Dates: Start 2020-01-15 (Actual); Primary Completion 2021-05-24 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pain intensity assessed by Visual Analogue Scale(VAS) | Baseline and Day 7
  Pain intensity is assessed by 100 mm Visual Analogue Scale(VAS) (0 mm = no pain and 100 mm = maximum pain) evaluated from baseline to Day 7.

SECONDARY OUTCOMES:
Change from baseline in pain intensity assessed by Visual Analogue Scale(VAS) | Baseline and Day 3
  Pain intensity is assessed by 100 mm Visual Analogue Scale(VAS) (0 mm = no pain and 100 mm = maximum pain) evaluated from baseline to Day 3.
Change from baseline in Finger to Floor Distance(FFD) | Baseline, Day 3 and Day 7
  FFD is measured by the Investigators who will ask the patients to bend forward and try to touch the floor with the fingers. The distance between the finger to the floor is measured in cm.
Change from baseline in Oswestry Disability Index(ODI) | Baseline, Day 3 and Day 7
  The questionnaire consists of 10 items with each item having 6 answers associated to activities of daily living. The ODI score range is 0 to 100% (low score: minimal disability, high score: bed-bound or exaggerating)
Change from baseline in Physician's Global Assessment of Response to Therapy(PGART) | Baseline and Day 7
  Physician's response of change after administration is assessed on 5-point rating scales(very poor, poor, no change, good and very good).

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hwan Moon, MD, Principal Investigator — Severance Hospital; Jin Hwan Kim, MD, Principal Investigator — Inje University; Tae Kyun Kim, MD, Principal Investigator — Wonkwang University Hospital
Locations (1):
- Navipharm, Suwon, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No